CLINICAL TRIAL: NCT02080104
Title: Intramuscular Versus Intravenous Prophylactic Oxytocin for the Third Stage of Labour Following Vaginal Delivery: A Randomised Controlled Trial
Brief Title: Intramuscular Versus Intravenous Prophylactic Oxytocin for Hemorrhage After Vaginal Delivery
Acronym: oxytocin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hediye Dagdeviren (Other Government)
Responsible Party: Sponsor-Investigator, Hediye Dagdeviren, md, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Organization: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27-01.14-02-02
Record Dates: First submitted 2014-03-01; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; oxytocin; vaginal delivery; prophylactic
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous 10 ıu oxytocin (Active Comparator): group which 2 ampul prophylactic oxytocin given for third stage of labour intravenously after vaginal delivery
  Interventions: Drug: intarvenous and intramusculer 10 IU oxytocin
- intramusculer 10 ıu oxytocin (Experimental): group which oxytocin administered intramusculary after vaginal delivery
  Interventions: Drug: intarvenous and intramusculer 10 IU oxytocin

INTERVENTIONS:
Drug: intarvenous and intramusculer 10 IU oxytocin — intarvenous and intramusculer 10 IU oxytocin

SUMMARY:
Intramuscular versus intravenous prophylactic oxytocin for the third stage of labour following vaginal delivery: A randomised controlled trial

DETAILED DESCRIPTION:
Prevention of postpartum haemorrhage is essential in the pursuit of improved health care for women. In this study investigators aimed to compare intramuscular oxytocin with intravenous oxytocin for the routine prevention of postpartum haemorrhage in women who deliver vaginally.In some countries, intravenous access can not be provided easily . Intramuscular application is faster , easier and tougher enforcement requires less skill and equipment . For this reason, less educated , which can be applied by those offering health services .

ELIGIBILITY:
Inclusion Criteria:

1. Research volunteers, the undersigned, pregnant women
2. Only with vaginal delivery (episiotomy and perineal tears can)
3. > 34 weeks or more will be
4. Cephalic presentation will be
5. At low risk of postpartum hemorrhage

Exclusion Criteria:

1. <18 years
2. Multiple pregnancies
3. The presence of uterine myoma
4. Having postpartum hemorrhage in previous pregnancies
5. Placenta previa, polyhydramnios
6. More than four parity
7. Fetal macrosomia
8. Hb <9mg/dl
9. preeclampsia
10. Uterine anomalies
11. Receiving anticoagulant therapy, suspected coagulopathy
12. > 42 weeks of pregnancy
13. Oxytocin allergy -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
early postpartum hemorrhage | postpartum 24 hours
  Blood loss during the birth and postpartum hemorrhage asset (within 24 hours> 500 cc blood loss)

SECONDARY OUTCOMES:
Blood transfusion requirement | postpartum 24 hours
  * Blood transfusion requirement
  * duration of phase 3 (> 30 min)
  * necessity of additional treatments for postpartum hemorrhage
  * the necessity of manual removal of placenta
  * side effects of the

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırkoy Dr Sadi Konuk Teaching and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Oladapo OT, Okusanya BO, Abalos E, Gallos ID, Papadopoulou A. Intravenous versus intramuscular prophylactic oxytocin for the third stage of labour. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD009332. doi: 10.1002/14651858.CD009332.pub4. PMID 33169839